CLINICAL TRIAL: NCT04218032
Title: Verenpaineen Seuranta Paineanturi-matriisilla
Brief Title: Wearable Blood Pressure Monitoring
Status: Completed | Type: Observational
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Matti Kaisti, Senior Research Fellow, University of Turku
Other Study IDs: 1574/31/2018
Record Dates: First submitted 2019-12-19; First posted 2020-01-06 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Blood Pressure
MeSH Terms: interventions — Sphygmomanometers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- blood pressure: blood pressure is measured from the participants, by using two methods. A new developed device and a reference device. The new device measures, using oscillometry, the blood pressure from the finger tip. The reference device is a standard sphygmomanometer.
  Interventions: Device: sphygmomanometer, SpyghmoCor, CNAP500

INTERVENTIONS:
Device: sphygmomanometer, SpyghmoCor, CNAP500 — blood pressure is measured with developed new non-invasive technology, oscillometry from the fingertip, and compared to non-invasive standard blood pressure measurement using a standard sphygmomanometer/SpyghmoCor device/CNAP500 device.

SUMMARY:
The goal of this study is to develop and validate a new non-invasive medical instrumentation technology for blood pressure measurement.

DETAILED DESCRIPTION:
The goal of this study is to develop and validate a new non-invasive medical instrumentation technology for assessing haemodynamic status measured from the fingertip using oscillometry. . As the finger pressing pressure is ramped up and then slowly down, an oscillometric response is recorded. From this signal the mean arterial pressure is found from which systolic and diastolic pressure is computed along with the full pressure waveform.

ELIGIBILITY:
Inclusion Criteria:

* written concent from the participant

Exclusion Criteria:

* pace maker, pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 33 volunteers (weight: mean 77 kg [range:48 to 117 kg]; height: mean 176 cm [range: 161 to 194 cm]; age: mean 32 [range: 23 to 75 years], 8 females) The subjects had a blood pressure range (DBP: 56 to 84 mmHg, SBP: 93 to 146 mmHg) and four of them were on blood pressure medication. Three measurements were performed on both the reference and the experimental device from which an average was calculated
  32 volunteers (age: mean 47 years [range: 24 to 83 years], 5 women). The validation study was carried out at Turku University Hospital. For reference manual auscultation was performed by two trained observers, and the maximum acceptable difference between the readings from the observers was 4 mmHg for both SBP and DBP. After an initial test measurement, three measurements were taken in a cyclical manner one device after another, both with the finger device and by auscultation.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Accuracy of new blood pressure measurement technology. | up to 12 weeks
  the accuracy of new developed blood pressure measurement technology is validated against existing gold standard method by comparing systolic and diastolic blood pressure values between the two.

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: No